CLINICAL TRIAL: NCT05989282
Title: Healthcare Organizational Structural Conditions and the Health of People Recently Released From Prison
Brief Title: Structural Conditions and Health After Release From Prison
Acronym: SCHARP
Status: Recruiting | Type: Observational
Sponsor: Kaiser Permanente (Other)
Collaborators: University of Colorado, Denver (Other); Denver Health and Hospital Authority (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB# 00002931; R01HL164106 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Diseases; Health Care Utilization
MeSH Terms: conditions — Cardiovascular Diseases; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exposure to structural conditions: Using a survey, we will measure participant exposure to organizational: access policies, transition programs, culture, support for social determinants of health and specialized services.

SUMMARY:
People released from prison experience two times higher cardiovascular (CV) mortality than the general population, have a high prevalence of poor CV health and increased risk of CV events within 2 years of release. Access to high quality healthcare following release from prison is key to preventing poor health and CV outcomes. Our study team will investigate facilitators and barriers to health care access experienced by people released from prison.

DETAILED DESCRIPTION:
Upon release from prison, people face numerous challenges including unstable housing, limited employment, stigma, and poor health. Structural conditions in healthcare systems, including policies, practices and attitudes around healthcare access, transition programs, culture, support of social determinants of health, and specialized services for people released from prison, may influence access and health outcomes for people released from prison. We will enroll people released from prison into a prospective cohort study to examine the association between exposure to structural conditions and 12-month primary outcomes of healthcare utilization (clinic visits, emergency visits, hospitalization) and secondary outcomes of CV hospitalization and all-cause mortality. Moderation by participant characteristics such as self-reported race, ethnicity, gender, age and baseline CV health will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Recenlty released from state prison into the Denver/Aurora Colorado metro area
* Age 18 and older
* Ability to understand study procedures in English or Spanish
* No plans to leave the area for six months

Exclusion Criteria:

* On "current inmate" status or still under correctional observation (i.e., under locked confinement part of the day or night)
* Plans to leave area within six months
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We are enrolling people who were formerly in prison. People on probation or on parole are responsible for meeting their own needs for health care, in contrast to people currently in prison, who receive these services from the prison system. Thus, people recently released from prison are a high-risk group for a range of poor health outcomes and poor access to care. For these reasons, the focus of this investigation is on people recently released from prison.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-05 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Healthcare utilization | 12 months
  Clinic visits, emergency visits, hospitalization

SECONDARY OUTCOMES:
Cardiovascular hospitalization | 12 months
  Hospitalization for a cardiovascular condition
Death | 12 months
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Daugherty, Principal Investigator — Kaiser Permanente Institute for Health Research
Locations (1):
- Kaiser Permanente Institute for Health Research, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No